CLINICAL TRIAL: NCT02021695
Title: DNA Methylation and Gene Expression in Qataris With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Other Study IDs: 13-00023 [JIRB]
Record Dates: First submitted 2013-11-22; First posted 2013-12-27 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: Non-diabetic controls: Group I: Non-diabetic controls Good overall health without history of Type II diabetes. Normal fasting glucose level (<100 mg/dL) and HbA1C < 5.7%
  Also:
  1. Must provide informed consent
  2. Males or Females aged 30 years or older to minimize the potential confounding of other forms of diabetes mellitus
  3. In patients with diabetes, no concomitant diseases except for micro- and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome (hypertension, dyslipidemia and obesity)
  4. Not taking any chronic medications (except of the diabetes and cardiovascular related drugs).
- Group II: Diabetic with HbA1C<7%: Group II:
  HbA1C<7%
  Also:
  1. Must provide informed consent
  2. Males or Females aged 30 years or older to minimize the potential confounding of other forms of diabetes mellitus
  3. In patients with diabetes, no concomitant diseases except for micro- and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome (hypertension, dyslipidemia and obesity)
  4. Not taking any chronic medications (except of the diabetes and cardiovascular related drugs).
- Group III: Good controlled diabetics with 7 % <HbA1C < 10%: Group III Good controlled diabetics with 7 % <HbA1C < 10%
  Also:
  1. Must provide informed consent
  2. Males or Females aged 30 years or older to minimize the potential confounding of other forms of diabetes mellitus
  3. In patients with diabetes, no concomitant diseases except for micro- and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome (hypertension, dyslipidemia and obesity)
  4. Not taking any chronic medications (except of the diabetes and cardiovascular related drugs).
- Group IV: Poorly controlled diabetics with HbA1C > 10%.: Group IV:
  Poorly controlled diabetics with HbA1C > 10%.
  Also:
  1. Must provide informed consent
  2. Males or Females aged 30 years or older to minimize the potential confounding of other forms of diabetes mellitus
  3. In patients with diabetes, no concomitant diseases except for micro- and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome (hypertension, dyslipidemia and obesity)
  4. Not taking any chronic medications (except of the diabetes and cardiovascular related drugs).

SUMMARY:
With the assessment of the healthy vs. diabetic and pre-diabetic Qatari population the investigators intend to measure the changes in DNA methylation and gene expression in blood monocytes and lymphocytes attributed to diabetes, and to evaluate whether theses changes are persistent or can be reversed by improving diabetes control.

DETAILED DESCRIPTION:
The global prevalence of Type 2 Diabetes (T2D) is rapidly rising throughout most regions of the developed and developing world. In Middle East countries, particularly in the Gulf Council countries, the diabetes pandemic along with the rates of obesity have risen due to the adoption of a modern lifestyle. In the Qatari population alone, T2D is highly prevalent as 18% of the Qatari adults are estimated to suffer from this disease. Consanguineous marriages, sedentary lifestyle, obesity and bad dietary habits are cited as the main causes for this high incidence rate. Chronic hyperglycemia caused by long-term uncontrolled diabetes state can lead to devastating complications such as cardiovascular diseases, neuropathy, and retinopathy. Such complications are also highly prevalent in the Qatari population, perhaps due to the relatively low adherence to clinical guidelines but vary among Qatari individuals based on their genetic predisposition and shared family environment.It is already known that inflammation is part of the complex biochemical process of initiating and further developing cardiovascular complications of diabetes. Experimental models have showed that exposure to hyperglycemia induces epigenomic changes in inflammatory pathways, which subsequently regulate gene expression leading to the development of vascular inflammation. The investigators therefore hypothesized that chronic hyperglycemia leads to altered DNA methylation and dysregulation of gene expression in peripheral blood monocytes and lymphocytes in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide informed consent
2. Males or Females aged 30 years or older to minimize the potential confounding of other forms of diabetes mellitus
3. In patients with diabetes, no concomitant diseases except for micro- and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome (hypertension, dyslipidemia and obesity)
4. Not taking any chronic medications (except of the diabetes and cardiovascular related drugs).

Exclusion Criteria:

1. Diagnosis of Type-I Diabetes
2. Active situational diabetes (steroids use/pregnancy)
3. Active infection or acute illness of any kind
4. Chronic inflammation (auto-immune diseases) or infection
5. Evidence of malignancy within the past 5 years
6. Chronic hematological disorders known to affect glycated hemoglobin results such as hemoglobinopathies (e.g. sickle cell disease and thalassemia), increases red-cell turnover (e.g. hemolytic anemia and spherocytosis.

   * Evidence of malignancy within the past 5 years
   * Chronic hematological disorders known to affect glycated hemoglobin results such as hemoglobinopathies

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited for the study at Hamad Medical Corporation. Most of the subjects will belong to the outpatients clinics. However, the subjects with bad Diabetes control might be recruited from the inpatient clinic as well.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2013-09; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
DNA methylation and gene expression in blood monocytes and lymphocytes | 1 hour
  Changes in DNA methylation and gene expression in blood monocytes and lymphocytes will be compared in healthy, diabetic and pre-diabetic subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Abi Khalil, MD, Principal Investigator — Weill Cornell Medical College in Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided